CLINICAL TRIAL: NCT04180800
Title: Studying the Association Between Folic Acid Deficiency and Social Isolation for Elderly Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7483
Record Dates: First submitted 2019-10-01; First posted 2019-11-29 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2019-10

CONDITIONS: Folic Acid Deficiency; Social Isolation; Elderly Patients
MeSH Terms: conditions — Folic Acid Deficiency; Social Isolation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Folic acid deficiency: Those with a folic acid defiency
  Interventions: Other: Lubben Social Network Scale - 6
- No deficiency: Those with no folic acid deficiency
  Interventions: Other: Lubben Social Network Scale - 6

INTERVENTIONS:
Other: Lubben Social Network Scale - 6 — One short oral interview to complete the Lubben Social Network Scale in auto-survey, translated in French. It contains 6 questions on 30 points, higher scores are associated with more social engagement, lower scores, specifically under 12/30, are associated with social isolation.

SUMMARY:
Social isolation among elderly people is a frequent and major determinant for health.

The risk of premature death is 2 to 5 time higher for socially isolated people, similarly for morbidity, duration of healing and complications rate.

Denutrition is also frequent for elderly people with potentially serious consequences. Vitamin deficiency, especially in B9 and B12 vitamins, are often associated with denutrition among elderly people.

Folic acid (vitamin B9) is not influenced by inflammation and folic acid income are necessarily exogene. Vitamin B9 is provided by fresh fruits and vegetables, and giblets.

The investigators observed a high prevalence in folic acid deficiency for socially isolated elderly patients. The investigators made the hypothesis that a folic acid defiency is associated with social isolation for elderly people.

The primary purpose is the study of the association between folic acid deficiency (measured by dosing of plasma concentration of vitamin B9) and social isolation evaluated by Lubben Social Network Scale in 6 questions.

The secondary purposes are the study of the correlation between folic acid deficiency and social conditions, nutritional status, biological data, poly pharmacy, cognitive functions, dependency and length of stay at hospital.

ELIGIBILITY:
Inclusion criteria :

* Patients hospitalized in geriatric rehabilitation care in Strasbourg University Hospital
* Age > 75 years
* Patient has given his consent

Exclusion criteria :

* Digestive malabsorption disorder : gastrectomy, extended intestinal resection, Crohn disease, celiac disease, parenteral nutrition
* Chronic alcoholism
* Treatment with sulfamids, methotrexate, anti epileptic treatment (hydantoin)
* Hemodialysis
* Patients under protection measure (curatorship, guardianship, judicial protection)
* Patient refuses to participate

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 75 years old, hospitalized in geriatric rehabilitation care in Strasbourg University Hospital
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
Measure of plasma concentration on vitamin B9 by blood test taken in regular hospital admission | 10 weeks
  Folic acid deficiency is evaluated by dosing of plasma concentration of vitamin B9 through blood test taken in regular hospital admission. Folic acid deficiency is defined by a concentration under 3 ng/mL.
Measure of social isolation by Lubben Social Network Scale in 6 questions | 10 weeks
  Social isolation is measured by score results on LSNS-6 auto-survey. A score lower than 12/30 is associated with social isolation.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine JEHL, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided